CLINICAL TRIAL: NCT02174510
Title: A Pharmacokinetic Study of Lurasidone After Single Oral Administration in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma (Suzhou) Co., Ltd. (Industry)
Collaborators: Xuhui Central Hospital, Shanghai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D1070002
Record Dates: First submitted 2014-02-11; First posted 2014-06-25 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2018-05

CONDITIONS: Schizophrenia
Keywords: pharmacokinetic; lurasidone; single dose
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 20mg lurasidone (Experimental): single oral lurasidone in 30 minutes after beginning of the over 350 kcal breakfast on day 1.The subjects will be follow up on day 8 to 11.
  Interventions: Drug: 20mg lurasidone; Drug: placebo
- 40mg lurasidone (Experimental): single oral lurasidone in 30 minutes after beginning of the over 350 kcal breakfast on day 1.The subjects will be follow up on day 8 to 11.
  Interventions: Drug: 40mg lurasidone; Drug: placebo
- 80mg lurasidone (Experimental): single oral lurasidone in 30 minutes after beginning of the over 350 kcal breakfast on day 1.The subjects will be follow up on day 8 to 11.
  Interventions: Drug: 80mg lurasidone; Drug: placebo

INTERVENTIONS:
Drug: 20mg lurasidone — single oral lurasidone or placebo in 30 minutes after beginning of the over 350 kcal breakfast on day 1.
  Arms: 20mg lurasidone
Drug: 40mg lurasidone — single oral lurasidone or placebo in 30 minutes after beginning of the over 350 kcal breakfast on day 1.
  Arms: 40mg lurasidone
Drug: 80mg lurasidone — single oral lurasidone or placebo in 30 minutes after beginning of the over 350 kcal breakfast on day 1.
  Arms: 80mg lurasidone
Drug: placebo

SUMMARY:
To evaluate the pharmacokinetic (PK) characteristics of lurasidone after single oral administration of different doses in healthy Chinese subjects.

To evaluate the safety and tolerability of lurasidone after single oral administration of different doses in healthy Chinese subjects.

DETAILED DESCRIPTION:
Single administration, double-blinded, placebo-controlled (3 subjects in each group will take placebo) and 3 dose groups (20 mg, 40 mg and 80 mg). There are three groups which are 20mg lurasidone or placebo, 40mg lurasidone or placebo and 80mg lurasidone or placebo.

This study comprises a screening period (between signing of the informed consent form and Day -2), baseline period (Day -1), treatment period (Days 1-3) and ending of study examination period (Days 8-11 after the last sample collection for PK evaluation).

ELIGIBILITY:
Inclusion Criteria:

1. After detailed explanations of study objectives, methods and procedures, anticipated efficacy, pharmacologic actions, risks and other relevant contents, subjects are aware of all relevant information related to this study and have signed the written informed consent form voluntarily.
2. Male subjects are 18≤ age <40 years of age when signing the informed consent.
3. Subjects with body weight of 50.0≤ and ≤ 80.0 kg and BMI (body mass index) of 19.0≤ and <24.0 at screening examination.
4. Subjects are able to comply with all requirements during this study period, receive various physical and laboratory examinations per study protocol, and report subjective symptoms.

Exclusion Criteria:

1. Based on the examination results during screening period, various physical and laboratory examinations performed 1 day before medication (Day-1 ) and before administration of study drug on the medication day, there are certain medical concerns on subject's health status in principal investigator's or study supervising physician's opinions (certain treatment or medical observation are deemed necessary).
2. Subjects with past diabetic history.
3. Subjects has an HbA1c level of >6.2% at screening.
4. Subjects with history of gastrointestinal operations.
5. Because of subjects' past medical history of cardiovascular diseases, liver diseases, renal diseases, endocrine disorders, digestive diseases, hematologic diseases, respiratory diseases, mental illness, neurological disorders (especially epilepsy and other convulsive disorders) and other diseases, subjects are unsuitable to participate in this study in the principal investigator's or study supervising physician's opinions.
6. Subjects with past history of allergy to drugs.
7. Subjects have consumed grapefruit or food containing grapefruit ingredients between 7 days before medication (Day -7) and administration of study drug on the medication day (Day 1). Subjects have consumed food containing hypericum perforatum L. ingredients between 14 days before medication (Day-14) and administration of study drug on the medication day (Day 1).
8. Subjects have taken any drugs (including over-the-counter drugs) between 7 days before medication (Day_-7) and administration of study drug on medication day.
9. Regular drinker (criteria are mean daily consumption ≥2 bottles of 640 mL beers or Chinese liquor≥150 mL).
10. Subjects are used to drink large amount (criteria are daily consumption>1.8 L) of caffeine-containing beverages (e.g. coffee, black tea, green tea, coca cola or nutritional oral solution, etc).
11. Subjects have history of drug abuse or positive urine drug tests.
12. Subjects with positive immunologic test results.
13. Average amount of daily smoking>20 cigarettes.
14. Subjects have taken other study drugs within 3 months (Day_-90~Day 1) before medication.
15. Subjects received lurasidone orally before.
16. Subjects have history of blood donations of 400 mL within 3 months (Day_-90~Day 1) before medication; 200 mL within 1 month (Day_-30~Day 1) before medication; or donation of blood components within 2 weeks (Day_-14~Day 1) before medication.
17. Subjects have consumed alcohol-containing food between 3 days before medication 3 (Day_-3) and before administration of study drug on medication day.
18. Subjects can not tolerate venipuncture or have poor peripheral venous access.
19. Subjects are unwilling to abstain from vigorous exercise from Day_-1 until discharge.
20. Other subjects who are unsuitable to participate in this study in principal investigator's or study supervising physician's opinions.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ChaoYing Hu, MD, Principal Investigator — Xuhui Center Hospital, Shanghai
Locations (1):
- Xuhui Center Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Hu C, Wang Y, Song R, Yu C, Luo X, Jia J. Single- and Multiple-Dose Pharmacokinetics, Safety and Tolerability of Lurasidone in Healthy Chinese Subjects. Clin Drug Investig. 2017 Sep;37(9):861-871. doi: 10.1007/s40261-017-0546-8. PMID 28695535

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 72 subjects were screened at the clinical site after obtaining informed consent. The data of informed consent from the first subject was march 2014. A total of 37 subjects were enrolled into the study and were randomized to three test drug groups (8 to 20mg group, 8 to 40mg group, 12 to 80mg group), and 9 subjects received placebo.
Groups:
- 20mg Lurasidone: 20mg lurasidone: single oral lurasidone.
- 40mg Lurasidone: 40mg lurasidone: single oral lurasidone.
- 80mg Lurasidone: 80mg lurasidone: single oral lurasidone.
- Placebo: Subjects administered placebo tablet at the same time with each lurasidone group.
Period: Overall Study
Arm/Group | 20mg Lurasidone | 40mg Lurasidone | 80mg Lurasidone | Placebo
Started | 8 | 8 | 12 | 9
Completed | 8 | 8 | 12 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study design included 28 men in the positive drug lurasidone group and 9 in placebo group. All subjects who received lurasidone or placebo were included in the safety population. All subjects who received lurasidone and have evaluable PK data were included in the PK analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | 20mg Lurasidone | 40mg Lurasidone | 80mg Lurasidone | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 12 | 9 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (3.74) | 25.4 (3.07) | 27.5 (7.79) | 28.4 (4.72) | 27.1 (5.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 8 | 8 | 12 | 9 | 37

OUTCOME MEASURES:

1. Primary Outcome: Lurasidone Cmax
Description: Cmax：Maximum (peak) observed drug serum concentration.
Time Frame: pre-dose,0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Population: ALL 28 subjects who received lurasidone and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | 20mg Lurasidone | 40mg Lurasidone | 80mg Lurasidone
Number analyzed (Participants) | 8 | 8 | 12
ng/ml | 32.9 (35.4) | 50.9 (29.6) | 113 (39.5)

2. Primary Outcome: Lurasidone AUC
Description: AUC：Area under the serum concentration-time curve
Time Frame: pre-dose,0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng･h/mL
Arm/Group | 20mg Lurasidone | 40mg Lurasidone | 80mg Lurasidone
Number analyzed (Participants) | 8 | 8 | 12
ng･h/mL
  AUC0-24 | 90.3 (26.3) | 151 (26.6) | 322 (34.8)
  AUC0-t | 97.9 (26.2) | 163 (26.5) | 353 (35.3)
  AUC0-∞ | 107 (26.3) | 174 (26.5) | 378 (35.6)

3. Primary Outcome: Lurasidone Tmax
Description: Tmax：Time to maximum (peak) drug serum concentration
Time Frame: pre-dose,0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Measure: Median (Full Range); unit: h
Arm/Group | 20mg Lurasidone | 40mg Lurasidone | 80mg Lurasidone
Number analyzed (Participants) | 8 | 8 | 12
h | 2.00 [1.0 to 2.0] | 2.00 [1.5 to 3.0] | 1.50 [1.0 to 2.0]

4. Primary Outcome: Lurasidone λZ
Description: λZ：Elimination rate constant
Time Frame: pre-dose,0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | 20mg Lurasidone | 40mg Lurasidone | 80mg Lurasidone
Number analyzed (Participants) | 8 | 8 | 12
1/h | 0.0271 (26) | 0.0383 (32.9) | 0.0383 (17.4)

5. Primary Outcome: Lurasidone t1/2
Description: t1/2 :Biological half life correlated with the elimination rate constant (kel) of semi-logarithmic concentration-time curve
Time Frame: pre-dose,0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | 20mg Lurasidone | 40mg Lurasidone | 80mg Lurasidone
Number analyzed (Participants) | 8 | 8 | 12
h | 25.5 (26) | 18.1 (32.9) | 18.1 (17.4)

6. Primary Outcome: Lurasidone MRT
Description: MRT：Mean residence time.
Time Frame: pre-dose,0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | 20mg Lurasidone | 40mg Lurasidone | 80mg Lurasidone
Number analyzed (Participants) | 8 | 8 | 12
h | 13.2 (26.3) | 11.1 (21.5) | 11.7 (13.7)

7. Primary Outcome: Lurasidone CL/F
Description: CL/F：Apparent total clearance.
Time Frame: pre-dose,0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | 20mg Lurasidone | 40mg Lurasidone | 80mg Lurasidone
Number analyzed (Participants) | 8 | 8 | 12
L/h | 187 (26.3) | 231 (26.5) | 212 (35.6)

8. Primary Outcome: Lurasidone VZ/F
Description: VZ/F: Apparent volume of distribution at terminal phase (correlated with λz)
Time Frame: pre-dose,0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | 20mg Lurasidone | 40mg Lurasidone | 80mg Lurasidone
Number analyzed (Participants) | 8 | 8 | 12
L | 6887 (36.3) | 6022 (41.8) | 5523 (39.0)

ADVERSE EVENTS:
Time Frame: From just after use of the study drug to the study-ending evaluation, up to 11 days.
Description: All 37 subjects who received lurasidone or placebo were included in the safety population.
Arm/Group | 20mg Lurasidone | 40mg Lurasidone | 80mg Lurasidone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 5/8 | 7/8 | 12/12 | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20mg Lurasidone (N=8) | 40mg Lurasidone (N=8) | 80mg Lurasidone (N=12) | Placebo (N=9)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood prolactin increased (Investigations) | 1 (1) | 1 (1) | 10 (10) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 5 (5) | 6 (6) | 12 (12) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other